CLINICAL TRIAL: NCT04837079
Title: National Survey of Essential Tremor Plus in China
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: NSETP-China
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Essential Tremor-plus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Clinical observational study — Clinical observational study

SUMMARY:
National Survey of Essential Tremor Plus in China（NSETP-China）is a multicenter cross-sectional study designed to investigate the clinical features of ET-plus in mainland China.

DETAILED DESCRIPTION:
Essential tremor (ET) is one of the most common adult-onset movement disorders, affecting 0.9% of the population across all ages worldwide. ET is a chronic, progressive neurologic disease whose the most recognizable clinical feature is a 4~12 Hz kinetic tremor of the upper limbs, usually occurring during a variety of voluntary movements. The etiology and pathogenesis of ET remain elusive.

Essential tremor-plus (ET-plus) is a new term coined in 2018 MDS consensus statement on tremor. ET-plus is defined as tremor with the characteristics of essential tremor, with additional neurological signs of uncertain clinical significance, such as impaired tandem gait, questionable dystonic posturing, memory impairment, or other mild neurological signs of unknown clinical significance that do not suffice to make an additional syndrome classification or diagnosis.

ET-plus is a controversial new concept. We will use scales or questionnaires to investigate the common soft neurological signs of ET-plus in mainland China. The details are as follows: (1) The tremor's impact on activities of daily living and clinical measurement of ET severity are evaluated by The Essential Tremor Rating Assessment Scale (TETRAS). (2) Cognitive condition is assessed by Mini Mental State Examination (MMSE) and Montreal Cognitive Assessment (MOCA). (3) The non-motor symptoms are evaluated by Non-motor Symptom Scale (NMSS). (4) Clinical assessment of balance and gait in ET-plus: we will use Tandem walk, Berg balance scale (BBS) and 10 meter walk timing test. (5) The Unified Dystonia Rating Scale (UDRS) for evaluation of dystonia in ET-plus. (6) The scale for the Assessment and Rating of Ataxia (SARA) is used to evaluate ataxia in ET-plus.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with ET and/or ET-plus by the Consensus Statement on the Classification of Tremors, from the Task Force on Tremor of the International Parkinson and Movement Disorder Society.

Exclusion Criteria:

Lack of capacity to consent to participate in the project

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients are Han Chinese from mainland China.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
The tremor's impact on activities of daily living and clinical measurement of ET severity are evaluated by The Essential Tremor Rating Assessment Scale (TETRAS). | May 1, 2021-April 30, 2022
  TETRAS consists of two subscales. The first one, Activities of Daily Living (ADL) Subscale contains 12 selfscored items, rating tremor's impact on ADL in a 0-4 Likert-type scale. Total score varies from 0-48. Higher score indicates a bigger impact on activities of daily living. The second part is the Performance Subscale, and is rated by clinicians'examination. The subscale is formed by 9 items that rate action tremor in the head, face, voice, limbs, and trunk from 0 to 4. Total score varies from 0-64. Higher score indicates severer tremor. For most items, the scores are defined only by whole numbers, but 0.5 increments may be used if you believe the rating is between two whole number ratings and cannot be reconciled to a whole number. Each 0.5 increment in rating is specifically defined for the assessment of upper limb postural and kinetic tremor and the dot approximation task (items 4 and 8).

SECONDARY OUTCOMES:
The non-motor symptoms are evaluated by Non-motor Symptom Scale. | May 1, 2021-April 30, 2022
  This scale includes 30 items which is divided into 9 domains. Total score varies from 0-360. Higher score indicates severer symptoms. Domain 1 evaluates cardiovascular system symptoms. Score of domain 1 varies from 0-24.
  Domain 2 evaluates sleep condition. Score of domain 2 varies from 0-48. Domain 3 evaluates cognitive function. Score of domain 3 varies from 0-72. Domain 4 evaluates illusion. Score of domain 4 varies from 0-36. Domain 5 evaluates attention and memory. Score of domain 5 varies from 0-36. Domain 6 evaluates gastrointestinal symptoms. Score of domain 6 varies from 0-36. Domain 7 evaluates urinary symptoms. Score of domain 7 varies from 0-36. Domain 8 evaluate sensory symptoms. Score of domain 8 varies from 0-24. Domain 9 evaluates other non-motor symptoms.
  Score of domain 9 varies from 0-48.
Cognitive condition is assessed by Mini Mental State Examination (MMSE). | May 1, 2021-April 30, 2022
  MMSE scale includes 30 items. Score of all the questions will be summed. All items were rated on a 2-point scale (0-1), with a minimal score of 0, and maximum total score of 30. A higher score demonstrates more better cognitive condition. The definition of cognitive disorder differs in education level. For those only receive elementary education, the cut-off value is 20. For other patients, presence of cognitive impairment was defined as MMSE scores less than 25.
Cognitive condition is assessed by Montreal Cognitive Assessment (MOCA). | May 1, 2021-April 30, 2022
  MOCA scale is a one page 30 point test. 16 items and 11 categories to assess multiple cognitive domains, including short-term memory recall task, visuospatial abilities, executive functions, attention, concentration and working memory, language and orientation to time and place. A cutoff 26 is used to define cognitive impairment. 1 point is added to the test-taker's score if they have 12 years education or less.
Tandem walk, Berg balance scale (BBS) and 10 meter walk timing test are used to evaluate balance and gait in ET-plus. | May 1, 2021-April 30, 2022
  Tandem walk：In this test, patients are asked to walk 10 steps on a straight path, with the heel of the leading foot touching the toe of the following foot. The number of missteps, defined as the number of steps away from the straight-line path, is the primary outcome reported. Balance is assessed by Berg Balance (BBS). The total score of the this scale is 56. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4. 0" indicates the lowest level of function and "4" the highest level of function. 0-20 on the BBS represents balance impairment; 21-40 on the BBS represents acceptable balance; 41-56 on the BBS represents good balance. Walking condition is assessed by 10 metre Walk Test (10 MWT). Patients walk without assistance 10 meters and the time is measured for the intermediate 6 meters to allow for acceleration and deceleration.
The Unified Dystonia Rating Scale (UDRS) for evaluation of dystonia in ET-plus. | May 1, 2021-April 30, 2022
  Dystonia postural is assessed by revised Dystonia Rating Scales (UDRS). The total score of this scale is 112, includes ratings for 7 items. For each of the items assessed, the UDRS has a severity and a duration rating. The severity rating is specific for each body region assessed and ranges from 0 (no dystonia) to 4 (extreme dystonia). The Duration rating assesses whether dystonia occurs at rest or with action, and whether it is predominantly at maximal or sub maximal intensity. The total score for the UDRS is the sum of the severity and duration factors.
The scale for the Assessment and Rating of Ataxia (SARA) is used to evaluate ataxia in ET-plus. | May 1, 2021-April 30, 2022
  SARA has eight items that yield a total score of 0 (no ataxia) to 40 (most severe ataxia); 1: gait (score 0 to 8), 2: stance (score 0 to 6), 3: sitting (score 0 to 4), 4: speech disturbance (score 0 to 6), 5: finger chase (score 0 to 4), 6: nose-finger test (score 0 to 4), 7: fast alternating hand movements (score 0 to 4), 8: heel-shin slide (score 0 to 4). Limb kinetic functions (items 5 to 8) are rated independently for both sides, and the arithmetic mean of both sides is included in the SARA total score.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China